CLINICAL TRIAL: NCT03799484
Title: Randomized, Single Center, Masked Study Comparing the Efficacy of Botulinum Toxin Type A Injection After Topical Anesthesia Versus Petrolatum Ointment
Brief Title: Botulinum Toxin Type A Injection After Topical Anesthesia Versus Petrolatum Ointment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Robert Cizik Eye Clinic (Other)
Responsible Party: Principal Investigator, Karina Richani-Reverol, Clinical Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HSC-MS-18-0908
Record Dates: First submitted 2019-01-03; First posted 2019-01-10 (Actual); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Forehead Rhytides; Forehead Wrinkles
Keywords: Rhytides; Forehead Wrinkles
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will only be known by the principal investigator performing the injections and will not be disclosed to the participants or the brow excursion examiner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Anesthesia (Other): 2.5% Lidocaine/2.5% Prilocaine Cream will be applied to one side of the forehead and Petrolatum Ointment to the other prior to administration of Botulinum Toxin Type A Injection
  Interventions: Drug: Botulinum toxin type A; Drug: 2.5% lidocaine/2.5% prilocaine
- Petrolatum (Other): Petrolatum Ointment will be applied to one side of the forehead and 2.5% Lidocaine/2.5% Prilocaine Cream to the other side prior to administration of Botulinum Toxin Type A Injection
  Interventions: Drug: Botulinum toxin type A; Device: petrolatum ointment

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin type A will be administered to both sides
  Other Names: BTX-A
Drug: 2.5% lidocaine/2.5% prilocaine — 2.5% lidocaine/2.5% prilocaine will be applied to one side of the forehead
  Other Names: EMLA
  Arms: Topical Anesthesia
Device: petrolatum ointment — petrolatum ointment will be applied to one side of the forehead
  Other Names: Aquaphor
  Arms: Petrolatum

SUMMARY:
The purpose of this study is to determine whether there is a difference in clinical effect, duration of effect, level of discomfort and patient satisfaction in patients receiving topical anesthesia on one side of the forehead and petrolatum ointment on the other prior to Botulinum Toxin Type A administration for the treatment of forehead rhytides.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-masked, comparative study in patients who present at the Robert Cizik Eye Clinic with horizontal forehead rhytides requiring treatment with botulinum toxin Type A (Botox ®; Allergan, Irvine, CA, USA).

The objective of this study is to determine whether there is a difference in clinical effect (weakness/paralysis of the frontalis muscle), duration of effect, level of discomfort and patient satisfaction in patients receiving topical anesthesia (2.5% lidocaine/2.5 % prilocaine cream, Impax Laboratories, LLC) on one side of the forehead and petrolatum ointment on the other prior to BTX-A administration for the treatment of forehead rhytides.

* Primary outcome variable is change of eyebrow excursion on each side of the forehead from baseline to each follow-up visit.
* Secondary outcome variables

  * Duration of effect, defined as the elapsed time from injection to the end of botulinum, such that return of baseline frontalis function, i.e. within 2 mm of baseline value
  * Perception of pain immediately after injection at each side
  * Patient satisfaction for each side
  * Patient's perception of difference in efficacy

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* Presence of horizontal forehead rhytides
* Good eyebrow excursion (greater than or equal to 5 mm)
* Able to understand and sign an informed consent form that has been approved by the Committee for the Protection of Human Subjects

Exclusion Criteria:

* Previous injection of botulinum toxin in the intended treatment area for the study within the last 4 months
* Known allergy to botulinum toxin
* Known history of sensitivity to local anesthetics of the amide type
* Existing disorder of neuromuscular transmission
* Usage of medication with effect on neuromuscular function
* Women of childbearing potential (who are not postmenopausal for at least 1 year or surgically sterile), who are pregnant or nursing or intend to become pregnant during the time of the study
* Significant brow asymmetry (> 5mm)
* Unable to follow-up for the duration of the study (16 weeks)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina Richani-Reverol, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Robert Cizik Eye Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott AB. Botulinum toxin injection into extraocular muscles as an alternative to strabismus surgery. J Pediatr Ophthalmol Strabismus. 1980 Jan-Feb;17(1):21-5. doi: 10.3928/0191-3913-19800101-06. PMID 7365644
- [Background] Carruthers A, Carruthers J. Clinical indications and injection technique for the cosmetic use of botulinum A exotoxin. Dermatol Surg. 1998 Nov;24(11):1189-94. doi: 10.1111/j.1524-4725.1998.tb04097.x. PMID 9834738
- [Background] Carter SR, Seiff SR. Cosmetic botulinum toxin injections. Int Ophthalmol Clin. 1997 Summer;37(3):69-79. doi: 10.1097/00004397-199703730-00006. No abstract available. PMID 9279643
- [Background] Charles PD. Botulinum neurotoxin serotype A: a clinical update on non-cosmetic uses. Am J Health Syst Pharm. 2004 Nov 15;61(22 Suppl 6):S11-23. doi: 10.1093/ajhp/61.suppl_6.S11. PMID 15598005
- [Background] Carruthers A, Carruthers J. Aesthetic indications for botulinum toxin injections. Plast Reconstr Surg. 1995 Feb;95(2):427-8. doi: 10.1097/00006534-199502000-00049. No abstract available. PMID 7824641
- [Background] Clark RP, Berris CE. Botulinum toxin: a treatment for facial asymmetry caused by facial nerve paralysis. Plast Reconstr Surg. 1989 Aug;84(2):353-5. PMID 2748749
- [Background] Sami MS, Soparkar CN, Patrinely JR, Hollier LM, Hollier LH. Efficacy of botulinum toxin type a after topical anesthesia. Ophthalmic Plast Reconstr Surg. 2006 Nov-Dec;22(6):448-52. doi: 10.1097/01.iop.0000248989.33572.3c. PMID 17117100
- [Background] Gordin EA, Luginbuhl AL, Ortlip T, Heffelfinger RN, Krein H. Subcutaneous vs intramuscular botulinum toxin: split-face randomized study. JAMA Facial Plast Surg. 2014 May-Jun;16(3):193-8. doi: 10.1001/jamafacial.2013.2458. PMID 24699554
- [Background] Li Y, Dong W, Wang M, Xu N. Investigation of the Efficacy and Safety of Topical Vibration Anesthesia to Reduce Pain From Cosmetic Botulinum Toxin A Injections in Chinese Patients: A Multicenter, Randomized, Self-Controlled Study. Dermatol Surg. 2017 Dec;43 Suppl 3:S329-S335. doi: 10.1097/DSS.0000000000001349. PMID 29016544
- [Background] Shi LL, Sargen MR, Chen SC, Arbiser JL, Pollack BP. Effective local anesthesia for onabotulinumtoxin A injections to treat hyperhidrosis associated with traumatic amputation. Dermatol Online J. 2016 Jun 15;22(6):13030/qt38b203d0. PMID 27617615
- [Background] Baumann LS, Grunebaum L, Elsaie ML, Murdock J, Jablonka E, Figueras K, Bell M. Safety and efficacy of a rapid-acting topical 4% lidocaine gel in a unique drug delivery system. J Drugs Dermatol. 2010 Dec;9(12):1500-4. PMID 21120257
- [Background] Weiss RA, Lavin PT. Reduction of pain and anxiety prior to botulinum toxin injections with a new topical anesthetic method. Ophthalmic Plast Reconstr Surg. 2009 May-Jun;25(3):173-7. doi: 10.1097/IOP.0b013e3181a145ca. PMID 19454924
- [Background] Alam M, Bolotin D, Carruthers J, Hexsel D, Lawrence N, Minkis K, Ross EV. Consensus statement regarding storage and reuse of previously reconstituted neuromodulators. Dermatol Surg. 2015 Mar;41(3):321-6. doi: 10.1097/DSS.0000000000000303. PMID 25705950
- [Background] Carruthers J, Fagien S, Matarasso SL; Botox Consensus Group. Consensus recommendations on the use of botulinum toxin type a in facial aesthetics. Plast Reconstr Surg. 2004 Nov;114(6 Suppl):1S-22S. doi: 10.1097/01.PRS.0000144795.76040.D3. PMID 15507786
- [Background] Ito H, Ito H, Nakano S, Kusaka H. Low-dose subcutaneous injection of botulinum toxin type A for facial synkinesis and hyperlacrimation. Acta Neurol Scand. 2007 Apr;115(4):271-4. doi: 10.1111/j.1600-0404.2006.00746.x. PMID 17376126
- [Background] Tzou CH, Giovanoli P, Ploner M, Frey M. Are there ethnic differences of facial movements between Europeans and Asians? Br J Plast Surg. 2005 Mar;58(2):183-95. doi: 10.1016/j.bjps.2004.10.014. PMID 15710113

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: 2.5% Lidocaine/2.5% Prilocaine Cream will be applied to one side of the forehead and Petrolatum Ointment to the other side of the forehead prior to administration of Botulinum Toxin Type A Injection.
Period: Overall Study
Arm/Group | All Participants
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Hispanic | 6
  White | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
Distance between both lateral canthi [Mean (Standard Deviation); unit: millimeters] | 98.29 (3.43)

OUTCOME MEASURES:

1. Primary Outcome: Eyebrow Excursion
Description: Participants will be asked to raise the brows, and the excursion of the brow from resting position to maximum elevation will be measured in millimeters.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: side of forehead (either left or right)
Arm/Group | Topical Anesthesia | Petrolatum
Number analyzed (Participants) | 14 | 14
Number analyzed (side of forehead (either left or right)) | 14 | 14
millimeters | 10.57 (3.3) | 10.57 (3.16)

2. Primary Outcome: Eyebrow Excursion
Description: as for outcome 1
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: side of forehead (either left or right)
Arm/Group | Topical Anesthesia | Petrolatum
Number analyzed (Participants) | 14 | 14
Number analyzed (side of forehead (either left or right)) | 14 | 14
millimeters | 3.46 (2.76) | 3.43 (2.93)

3. Primary Outcome: Eyebrow Excursion
Description: as for outcome 1
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: side of forehead (either left or right)
Arm/Group | Topical Anesthesia | Petrolatum
Number analyzed (Participants) | 14 | 14
Number analyzed (side of forehead (either left or right)) | 14 | 14
millimeters | 5.96 (2.62) | 5.68 (2.55)

4. Primary Outcome: Eyebrow Excursion
Time Frame: week 16
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: side of forehead (either left or right)
Arm/Group | Topical Anesthesia | Petrolatum
Number analyzed (Participants) | 14 | 14
Number analyzed (side of forehead (either left or right)) | 14 | 14
millimeters | 8.21 (2.89) | 8.07 (2.97)

5. Secondary Outcome: Duration of Botulinum Toxin Type A Effect
Description: Loss of Botulinum Toxin Type A effect is defined as return of baseline frontalis muscle function (function prior to injection) as indicated by eyebrow excursion measurement within 2 millimeters of baseline value.
Time Frame: week 16
Measure: Mean (Standard Error); unit: weeks
Units Other Than Participants: side of forehead (either left or right)
Arm/Group | Topical Anesthesia | Petrolatum
Number analyzed (Participants) | 14 | 14
Number analyzed (side of forehead (either left or right)) | 14 | 14
weeks | 14.2857 (1.2317) | 15.2857 (0.7301)

6. Secondary Outcome: Perception of Pain Immediately After Injection as Assessed by a Visual Analogue Scale
Description: A visual analogue scale will be used to assess pain. The scale ranges from 0 (no pain) to 10 (the worse pain possible), with lower scores indicating a better outcome.
Time Frame: Immediately after botox injection
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: side of forehead (either left or right)
Arm/Group | Topical Anesthesia | Petrolatum
Number analyzed (Participants) | 14 | 14
Number analyzed (side of forehead (either left or right)) | 14 | 14
units on a scale | 2.43 (1.55) | 3.96 (1.74)

7. Secondary Outcome: Participant Satisfaction With Overall Appearance of Forehead as Assessed by a Patient Satisfaction Survey
Description: The survey will be assessed using a rating scale with the following categories: very satisfied, satisfied, neutral, dissatisfied, and very dissatisfied.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  very satisfied | 8
  satisfied | 6
  neutral | 0
  dissatisfied | 0
  very dissatisfied | 0

8. Secondary Outcome: Participant Satisfaction With Overall Appearance of Forehead as Assessed by a Patient Satisfaction Survey
Description: as for outcome 7
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  very satisfied | 7
  satisfied | 6
  neutral | 1
  dissatisfied | 0
  very dissatisfied | 0

9. Secondary Outcome: Participant Satisfaction With Overall Appearance of Forehead as Assessed by a Patient Satisfaction Survey
Description: as for outcome 7
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  very satisfied | 8
  satisfied | 2
  neutral | 1
  dissatisfied | 3
  very dissatisfied | 0

10. Secondary Outcome: Participant Satisfaction With Appearance of Right Side of Forehead as Assessed by a Patient Satisfaction Survey
Description: as for outcome 7
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  very satisfied | 8
  satisfied | 6
  neutral | 0
  dissatisfied | 0
  very dissatisfied | 0

11. Secondary Outcome: Participant Satisfaction With Appearance of Right Side of Forehead as Assessed by a Patient Satisfaction Survey
Description: as for outcome 7
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  very satisfied | 7
  satisfied | 5
  neutral | 2
  dissatisfied | 0
  very dissatisfied | 0

12. Secondary Outcome: Participant Satisfaction With Appearance of Right Side of Forehead as Assessed by a Patient Satisfaction Survey
Description: as for outcome 7
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  very satisfied | 8
  satisfied | 2
  neutral | 1
  dissatisfied | 3
  very dissatisfied | 0

13. Secondary Outcome: Participant Satisfaction With Appearance of Left Side of Forehead as Assessed by a Patient Satisfaction Survey
Description: as for outcome 7
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  very satisfied | 8
  satisfied | 6
  neutral | 0
  dissatisfied | 0
  very dissatisfied | 0

14. Secondary Outcome: Participant Satisfaction With Appearance of Left Side of Forehead as Assessed by a Patient Satisfaction Survey
Description: as for outcome 7
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  very satisfied | 6
  satisfied | 7
  neutral | 1
  dissatisfied | 0
  very dissatisfied | 0

15. Secondary Outcome: Participant Satisfaction With Appearance of Left Side of Forehead as Assessed by a Patient Satisfaction Survey
Description: as for outcome 7
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants
  very satisfied | 8
  satisfied | 2
  neutral | 1
  dissatisfied | 3
  very dissatisfied | 0

16. Secondary Outcome: Number of Participants Who Perceive a Difference in Efficacy Between the 2 Sides of Their Face
Description: Participants will be asked if there is a noticeable difference between the 2 sides of their face.
Time Frame: Week 2
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants | 3

17. Secondary Outcome: Number of Participants Who Perceive a Difference in Efficacy Between the 2 Sides of Their Face
Description: Participants will be asked if there is a noticeable difference between the 2 sides of their face.
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants | 2

18. Secondary Outcome: Number of Participants Who Perceive a Difference in Efficacy Between the 2 Sides of Their Face
Description: Participants will be asked if there is a noticeable difference between the 2 sides of their face.
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Topical Anesthesia | Petrolatum
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT03799484/Prot_SAP_000.pdf